CLINICAL TRIAL: NCT02888704
Title: Phase I Clinical Trial to Evaluate the Safety, Tolerance, and Exploratory Efficacy of ADSTEM Inj. in Patients With Moderate to Severe, Subacute and Chronic Atopic Dermatitis
Brief Title: Safety and Efficacy of ADSTEM Inj. in Patients With Moderately Subacute and Chronic Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EHL Bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AD-CP-15-1; 30902 (Other Grant/Funding Number: Republic or Korea Ministry of Food and Drug Safety)
Record Dates: First submitted 2016-08-15; First posted 2016-09-05 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Mesenchymal stem cells
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention: Biological: ADSTEM Inj. (Experimental): 1. ADSTEM Inj. 1.0x10^8 mesenchymal stem cells as an intravenous infusion once for the duration of the study.
  2. ADSTEM Inj. 3.0x10^8 mesenchymal stem cells as an intravenous infusion once for the duration of the study.
  Interventions: Drug: ADSTEM Inj. (Adult human mesenchymal stem cells)

INTERVENTIONS:
Drug: ADSTEM Inj. (Adult human mesenchymal stem cells) — Comparison of different dosages of the drug in the aspect of safety and efficacy.
  Other Names: ADSTEM Inj.

SUMMARY:
This study aims to evaluate safety, tolerance, and efficacy in subjects with over moderately subacute and chronic atopic dermatitis after an intravenous injection of autologous mesenchymal stem cells. The study is composed of two steps. Step 1 is to determine clinically proper dose capacity of the ADSTEM Inj. and step 2 is to evaluate exploratory efficacy of the ADSTEM Inj. at the proper dose.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a type of inflammation of the skin. It results in itchy, swollen, red, and cracked skin. The symptoms typically start in childhood with changing severity over the years. The pathogenesis of AD is characterized by excessive type 2 helper T cell mediated inflammatory responses, resulting in B lymphocyte mediated increase in serum level of immunoglobulin E (IgE). Subsequent degranulation of mast cells by IgE releases various inflammatory mediators, which recruit the lymphocytes and eosinophils into the lesion.

Current clinical management of AD includes topical corticosteroids and systemic immunosuppressants. However, these drugs have been reported to carry the risk of side-effects and severe.

Several recent studies including ours have demonstrated that mesenchymal stem cells (MSCs) could suppress allergic responses in AD. MSCs have been known to interact with cell types of both innate and adaptive immune systems, which results in the suppressive effect on proliferation, differentiation, and activation of immune cells including T cells, B cells, dendritic cells, and natural killer cells. Indeed, a number of studies have reported that the immunomodulatory ability of MSCs can be usefully applied for the treatment of autoimmune and inflammation-related diseases such as asthma, rhinitis, and dermatitis. Therefore, MSCs has possibility as a new drug for AD.

ELIGIBILITY:
Inclusion Criteria:

* Of either gender, aged ≥19 and ≤70 years
* Atopic dermatitis subjects who are coincident with Hanifin and Rajka diagnosis criteria
* Subacute and chronic atopic subjects who have atopic dermatitis symptoms continually at least 6 months
* Subjects with over moderate atopic dermatitis (SCORAD score > 20)
* Subjects who understand and voluntarily sign an informed consent form

Exclusion Criteria:

* Subjects who have systemic infection
* Subjects who have human Immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV)
* Subjects who need to take the medicine which is prohibited during this study
* Subjects who have asthma
* Subjects who can not stop treatment with topical steroids (group 1~5), oral antibiotics, whole body photochemotherapy, immunosuppressive drug within 4 weeks before the treatment visit
* Pregnant, breast-feeding women or women who plan to become pregnant during this study (Females of childbearing potential must have a negative urine pregnancy test)
* Subjects who currently participate in other clinical trial or participated in other clinical trial within 30 days
* Subjects who had a serious adverse events during stem cell therapy
* Subjects who had a hypersensitivity to antibiotics or antimycotics
* Subjects who creatinine value is more than two times of the upper limit of the normal range at screening test
* Subjects who aspartate transaminase/alkaline transaminase (AST/ALT) value is more than three times of the upper limit of the normal range at screening test
* Subjects who have any other condition which the investigator judges would make patients unsuitable for study participation

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The number of subjects with treatment-related adverse events as assessed by CTCAE version 4.03 | 12 weeks follow-up after treatment
  physical exam, vital sign, laboratory findings, and adverse drug reactions

SECONDARY OUTCOMES:
The reduction ratio of scoring atopic dermatitis (SCORAD) index as contrasted with baseline value | 12 weeks follow-up after treatment
The variation of SCORAD index as contrasted with baseline value | 12 weeks follow-up after treatment
The variation of each index score of SCORAD index as contrasted with baseline value | 12 weeks follow-up after treatment
  TBSA, erythema, edema/papulation, oozing/crusting, excoriation, lichenification, dryness, pruritus, and insomnia
The variation of the degrees of disease as contrasted with baseline value | 12 weeks follow-up after treatment
The variation of investigator's global assessment (IGA) as contrasted with baseline value | 12 weeks follow-up after treatment
The variation of eczema area and severity index (EASI) total score as contrasted with baseline value | 12 weeks follow-up after treatment
The variation of total immunoglobulin E (IgE) in serum as contrasted with baseline value | 12 weeks follow-up after treatment
The variation of total prostaglandin E2 (PGE2) in serum as contrasted with baseline value | 12 weeks follow-up after treatment
The variation of total eosinophil cationic protein (ECP) in serum as contrasted with baseline value | 12 weeks follow-up after treatment
The variation of total Chemokine ligand 17 (CCL17) in serum as contrasted with baseline value | 12 weeks follow-up after treatment
The variation of total Chemokine ligand 27 (CCL27) in serum as contrasted with baseline value | 12 weeks follow-up after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Young-joon Seo, M.D., Ph.D, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, Chungcheongnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No